CLINICAL TRIAL: NCT05976542
Title: Investigation of the Relationship Between Plantar Fascia and Achilles Tendon Thickness Asymmetry and Spatio-temporal Parameters of Gait in Healthy Individuals
Brief Title: The Relationship Between Plantar Fascia and Achilles Tendon Thickness Asymmetry and Spatio-temporal Parameters of Gait
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Pınar Kısacık, PhD, Principle Investigator, Hacettepe University
Other Study IDs: GO 23/442
Record Dates: First submitted 2023-07-19; First posted 2023-08-04 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Achilles Tendon Thickness; Plantar Fascia Thickness; Spatio-temporal Parameteres of Gait
Keywords: Achilles tendon thickness; Plantar fascia thickness; Spatio-temporal parameteres of gait

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There are studies on loading the foot with an increase in the thickness of the Plantar Fascia and Achilles Tendon.

However, no study was found that evaluated the relationship between morphological features such as plantar fascia and Achilles tendon thickness and spatio-temporal parameters of gait in healthy individuals.

In this study, it is aimed to investigate the relationship between the asymmetry in the thickness of the plantar fascia and Achilles tendon and the asymmetry in the spati-temporal parameters of gait.

Healthy adult volunteers aged 20-40 will participate in the research. Demographic data of the participants will be recorded in the study. Following this, a clinical evaluation of the foot and ankle will be made. The Optogait Photoelectric Cell System (Microgate, Bolzano, Italy) device will be used to record the spatio-temporal parameters of gait, and the Sonostar Double Head Wireless Mini Ultrasound device (Sonostar Inc., China) will be used to assess the thickness of the plantar fascia and Achilles tendons.

ELIGIBILITY:
Inclusion Criteria:

* Being physically healthy (No symptoms or complaints at the moment, and no disease or trauma affecting the musculoskeletal system in the last 6 months)
* Being 20-40 years old
* Body Mass Index (BMI) being within the limits accepted as normal (18.5-24.9kg/m2) according to the World Health Organization (WHO)
* Classification of foot type as normal (API score= 0 to +5) as a result of the evaluation made with the Foot Posture Index (API) (38)
* Not having done any compelling (jogging, walking, weight or resistance training, yoga, pilates, aerobics, collective exercise sessions such as stepping…) exercises and activities in the last 2 days before the evaluation.

Exclusion Criteria:

* Disease or problems that may affect walking (plantar fasciitis, having to use walking aids, visual or hearing impairment, other problems related to the lower extremities or spine)
* Having undergone orthopedic trauma or surgery involving the lower extremity
* Having symptoms of severe shortness of breath or intolerance of walking while walking
* Person; have a medical history that may indicate an increased risk of falling, such as fainting of unknown cause, blood sugar imbalance, unstable low or high blood pressure
* Congenital (pes planus, pes cavus, pes equinovarus, vertical talus, etc.) or acquired (pes planus and planovalgus, pes cavus, other deformities associated with foot arches…) foot deformity defined by clinical evaluation
* Presence of cardiovascular, neurological or musculoskeletal orthopedic or rheumatological disease or systemic disease associated with diabetes, connective tissue disorder
* In addition, hypoechoic areas, perifascial fluid, and plantar fascia thickness measuring more than 4 mm during ultrasound imaging (39).

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult volunteers aged 20-40 will participate in the research.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-05 (Estimated)

PRIMARY OUTCOMES:
Plantar fascia thickness | Day 1
  One of the researcher measured the thickness of the plantar fascia using Clarius L7 linear ultrasound. To image the plantar fascia, we positioned the patient in the prone position with the feet hanging off the table and the subtalar joint stabilized in the neutral position. Here, we placed the ultrasound probe on the line between the medial condyle of the calcaneus and the 2nd and 3rd toes and clearly showed the calcaneus.
Achilless tendon thickness | Day 1
  One of the researcher measured the thickness of the Achilles tendon using Clarius L7 linear ultrasound. To image the Achilles tendon, we positioned the patient in the prone position with the feet hanging off the table and the subtalar joint stabilized in the neutral position. We measured the thickness of the tendon both longitudinally and transversely from the projection of the medial malleolus to the posterior aspect. We applied plenty and sufficient amount of gel to minimize the pressure and increase the contact and took 3 repeated images. We made an effort to minimize the pressure as much as possible during image acquisition.
Spatio-temporal parameters of gait | Day 1
  The OptoGait Photoelectric Cell System (Microgate, Bolzano, BZ, Italy) was used to set up for collecting spatiotemporal parameters of gait and was calibrated by the manufacturer. The system was linked via an interface unit to a computer and the OptoGait software program (Microgate, Bolzano, Italy) used. The following spatiotemporal parameter of gait were extracted: step length (cm), stance phase (percent of gait cycle [%GC]), swing phase (%GC), single support (%GC), loading response (%GC), preswing (%GC), and step time (s), stride length (cm), double support (%GC), stride time (sec), cadence (steps/min), and gait speed (m/sec).
  For familiarization of participants to treadmill, 6-minute trial-session used based on the study of Meyer et al (Meyer et al., 2019). For the test protocol; participants were asked to walk at self-selected walking pace for 1 minute on barefoot.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Kısacık, Principal Investigator — Hacettepe University

IPD SHARING:
Plan to Share IPD: No